CLINICAL TRIAL: NCT04471818
Title: Ketamine Versus Placebo as Adjuvant Treatment for Major Depressive Disorder and Wish to Hasten Death in Advanced Cancer Patients Undergoing Palliative Care
Brief Title: Ketamine or Placebo in Patients With Major Depression and Advanced Cancer
Acronym: KODIAC
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Instituto Nacional de Cancerologia de Mexico (Other)
Responsible Party: Principal Investigator, Oscar Raúl Rodríguez Mayoral, Head psychiatrist at the Palliative Care Unit of the National Cancer Institute (INCan, Mexico), Instituto Nacional de Cancerologia de Mexico
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: (019/024/CPI) /CEI/1332/18)
Record Dates: First submitted 2020-06-16; First posted 2020-07-15 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Major Depressive Disorder; Advanced Cancer
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketamine (Experimental): Patients allocated to the ketamine arm will receive 0.5 mg/kg of ketamine every week administered intravenously for 4 weeks.
  Interventions: Drug: Ketamine
- Placebo (Placebo Comparator): Patients allocated to the ketamine arm will receive 0.5 mg/kg of ketamine every week administered intravenously for 4 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Ketamine — Ketamine (0.5 mg/kg) will be administered intravenously once every week to patients in the experimental arm of the study
  Arms: Ketamine
Other: Placebo — Placebo (0.5 mg/kg) will be administered intravenously once every week to patients in the experimental arm of the study
  Arms: Placebo

SUMMARY:
Major depression (MD) is a psychiatric disorder characterized by a persistent feeling of sadness, anhedonia or a decreased perception of pleasurable experiences, as well as appetite alterations and weight variations, sleep disorders, altered psychomotor skills, fatigue, guilt, decreased self-worth, suicidal thoughts and difficulty concentrating in a task (1).

MD is a frequent complication in patients who are diagnosed with advanced cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 to 65 years of age
2. Sex: Male or female
3. Major depressive disorder (MDD) diagnosis as per Diagnostic and Statistical Manual of Mental Disorders (DSM-5).
4. Palliative stage cancer diagnosis (advanced-disease stage)
5. Who can read and write in spanish
6. Eastern Cooperative Oncology Group (ECOG) 0-2
7. Karnofsky ≥ 50
8. Palliative prognostic index A
9. Not currently undergoing systemic oncologic treatment
10. Patients who agree to participate in the study by signing an informed consent.

Exclusion Criteria:

1. Comorbidities including other psychiatric diseases (additional to MDD, generalized anxiety or panic disorder).
2. Magnetic resonance or computerized tomography with major structural alterations.
3. Pregnant or breastfeeding women.
4. Patients with hypersensitivity to ketamine
5. Cardiac insufficiency
6. Patients with a history of psychosis
7. Patients with first-degree relatives with a history of psychosis
8. Patients with uncontrolled glaucoma
9. Current neurological illness

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2019-09-19 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Brief Edinburg Depression Scale (BEDS) score | 3 weeks
  Scale to assess depression validated in cancer patients. For the BEDS scale, 6 items are included and scored, maximum score is 18 and minimum score is 0. Patients screened for depression are considered cases when scoring ≥7 in this scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Nacional de Cancerología (INCan), Mexico City, Mexico